CLINICAL TRIAL: NCT03794843
Title: A Randomized, Open-label, Single Dose, Two Formulation, Two Period, Double Cross Over Bioavailability Comparison Study of Two Types of Nimodipine Injections in Healthy Volunteers
Brief Title: Bioavailability Comparison Study of Two Types of Nimodipine Injections in Healthy Volunteers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenyang Dongxing Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BJK-PK-NMDP-201801
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Bioavailability; Safety Issues; Ischemic Cerebrovascular Disease
Keywords: Nimodipine; bioavailability; Safety; ischemic cerebrovascular disease
MeSH Terms: interventions — Nimodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nimodipine Injection (II) (Experimental): The specification of this injection is 5 ml: 4 mg , which is administered by constant infusion intravenously with an infusion pump. The injection and 0.9% sodium chloride injection is simultaneously infused at a ratio of 1:16 (injection: combined infusion). The rate of intravenous drip was started at 0.5 mg/h for 2 hours, and the rate of intravenous drip was 1.0 mg/h after 2 hours, and continuous infusion for 12 hours, for a total of 11 mg of nimodipine.
  Interventions: Drug: Nimodipine Injection (II)
- Nimodipine Injection (Experimental): The specification of this injection is 50 ml: 10 mg ,which is administered by constant infusion intravenously with an infusion pump. The injection and 0.9% sodium chloride injection is simultaneously infused at a ratio of 1:4 (injection: combined infusion). The rate of intravenous drip was started at 0.5 mg/h for 2 hours, and the rate of intravenous drip was 1.0 mg/h after 2 hours, and continuous infusion for 12 hours, for a total of 11 mg of nimodipine.
  Interventions: Drug: Nimodipine Injection

INTERVENTIONS:
Drug: Nimodipine Injection — Nimodipine injection (trade name: Nimotop) manufactured by Bayer Pharma AG was used as the reference preparation
  Other Names: Nimotop
  Arms: Nimodipine Injection
Drug: Nimodipine Injection (II) — Nimodipine Injection (II) was supplied by Shenyang Dongxing Pharmaceutical Technology Co., Ltd
  Arms: Nimodipine Injection (II)

SUMMARY:
A Randomized, Open-label, Single Dose, Two Formulation, Two Period, Double Cross Over Bioavailability Comparison Study of two types of Nimodipine Injections in Healthy Volunteers.

DETAILED DESCRIPTION:
The investigation product Nimodipine Injection (II) was supplied by Shenyang Dongxing Pharmaceutical Technology Co., Ltd.And Nimodipine injection (trade name: Nimotop) manufactured by Bayer Pharma AG was used as the reference preparation.The volunteers were administered with Nimodipine injection for intravenous infusion (containing nimodipine 11 mg) for 12 consecutive hours, respectively.The Venous blood was collected at 0 hours before the administration (ie, 1 hour before the administration) and 10 minutes, 20 minutes, 30 minutes, 45 minutes, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12 h (Administration was over) and 12.5 h, 13 h, 14 h, 16 h, 19 h, 22 h, 25 h, 36 h, 3 ml per blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the study, and fully understand the test content, process and possible adverse reactions, and be able to comply with the protocol according to the test plan requirements;
2. Healthy subjects, both male and female;
3. Age ≥ 18 years old;
4. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index in the range of 19 ~ 26 (including the critical value)[Body mass index (BMI) = weight (kg) / height 2 (m2)].

Exclusion Criteria:

- Subject who is in one of the following conditions may not be eligible.

1. Those who smoke more than 5 cigarettes per day for 3 months before the test or who cannot stop smoking during the trial period;
2. Allergies, such as those who are allergic to drugs, food and pollen, or those known to be allergic to nimodipine;
3. Those who have a history of alcohol abuse 6 months before the test (defined as drinking 14 units of alcohol per week: 1 unit = 285 ml of beer, or high-alcohol (50% or more alcohol) 25 ml, or 150 ml of wine) or Drinkers cannot be stopped during the trial;
4. Donor blood or a large amount of blood loss ≥400 ml (excluding female menstrual blood volume) within 3 months before the test, or have a history of halo and fainting;
5. Anyone taking any drug within 14 days before the test;
6. Antidepressants (such as fluoxetine), nortriptyline, norfloxacin, anti-HIV drugs (such as azidothymidine), calcium antagonists (such as nifedipine), were used within 28 days prior to the test. Diltiazem, verapamil, alpha-methyldopa and other antihypertensive drugs;
7. Have taken the study drug within 3 months before the test, or participated in any drug or medical device clinical trial;
8. Clinical laboratory examination, vital signs, physical examination, and 12-lead ECG abnormalities in the screening period are clinically significant;
9. During screening, when staying in the clinical center, the supine pressure of the supine position is not in the range of 100~139 mmHg, and the diastolic pressure in the supine position is not in the range of 60~89 mmHg;
10. During screening, when staying in the clinical center, the pulse is not in the range of 60~100 beats/min before each dose;
11. There is a serious arrhythmia: QTc interval prolongation (QTc over 450 ms), or QTc interval prolongation syndrome or family history of sudden death
12. A positive result of screening for hepatitis B surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody or Treponema pallidum-specific antibody;
13. Health status: a history of major diseases or important organ diseases such as nervous system, mental system, respiratory system, cardiovascular system, digestive system, blood system, endocrine system, musculoskeletal or metabolic abnormalities;
14. pregnant and lactating women;
15. Female subjects of childbearing age have a pregnancy plan or unable to take effective contraception after the first dose and within 3 months after the last dose, from 30 days before screening to 3 months after the last dose. Measures (non-pharmaceutical contraception), see the appendix for specific contraceptive measures;
16. Can not stop taking chocolate, any caffeinated food or drink during the test; or eat any food or drink containing grapefruit ingredients 14 days before the first dose to the end of the test;
17. Those who are positive for alcohol screening before dosing, or who have taken any alcoholic products within 24 hours prior to dosing;
18. Those who are positive for drug screening, who have had a history of drug abuse in the past five years or who have used drugs three months before the trial;
19. Investigators believe that it is not appropriate to participate in this test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
AUC | Within 36 hours after starting the administration
  Evaluation of bioequivalence based on pharmacokinetic parameters such as AUC
Cmax | Within 36 hours after starting the administration
  Evaluation of bioequivalence based on pharmacokinetic parameters such as Cmax

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No